CLINICAL TRIAL: NCT02353754
Title: A Multicenter, Open-Label Study to Evaluate the Safety and Efficacy of EXPAREL When Administered Via Infiltration Into the Transversus Abdominis Plane (TAP) After Bupivacaine Spinal Anesthesia in Subjects Undergoing Elective Cesarean Section
Brief Title: Evaluation of the Safety and Efficacy of EXPAREL When Administered Into the TAP in Subjects Undergoing Cesarean Section
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment. None of the subjects received EXPAREL.
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-402
Record Dates: First submitted 2015-01-28; First posted 2015-02-03 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Subjects in Group 1 (Standard of Care) will receive intrathecal morphine injection (e.g., Duramorph®) 0.2 mg in conjunction with the single-shot spinal anesthesia. No TAP block will be administered.
  Interventions: Drug: Intrathecal morphine injection
- EXPAREL/TAP (Experimental): Subjects in Group 2 will receive a bilateral TAP infiltration with a single 20 mL dose of EXPAREL 266 mg expanded in volume with 20 mL of normal saline for a total volume of 40 mL (20 mL infiltrated on each side of the abdomen).
  Interventions: Drug: EXPAREL

INTERVENTIONS:
Drug: Intrathecal morphine injection — 0.2 mg
  Other Names: Duramorph
  Arms: Standard of Care
Drug: EXPAREL — 266 mg
  Other Names: Bupivacaine liposome injectable suspension
  Arms: EXPAREL/TAP

SUMMARY:
This is a Phase 4, multicenter, open-label study evaluating EXPAREL infiltration into the transversus abdominis plane (TAP) after bupivacaine hydrochloride (HCl) spinal anesthesia in subjects undergoing elective Cesarean section (C-section).

DETAILED DESCRIPTION:
There will be two groups of subjects with approximately 40 subjects per group. Prior to the C-section, all subjects will receive single-shot spinal anesthesia (1.5 mL bupivacaine HCl 0.75% with dextrose 8.25%). Subjects in Group 1 (Standard of Care) will receive intrathecal morphine injection (e.g., Duramorph®) 0.2 mg in conjunction with the single-shot spinal anesthesia. No TAP block will be administered. Subjects in Group 2 (EXPAREL/TAP) will receive a bilateral TAP infiltration with a single 20 mL dose of EXPAREL 266 mg expanded in volume with 20 mL of normal saline for a total volume of 40 mL (20 mL infiltrated on each side of the abdomen).

ELIGIBILITY:
Inclusion Criteria:

1. Females ≥18 years of age at screening.
2. Scheduled to undergo elective C-section (single or multiple births).
3. American Society of Anesthesiology (ASA) physical status 1, 2, or 3.
4. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics or opioids.
2. Contraindication to bupivacaine, morphine, ketorolac, ibuprofen, or acetaminophen.
3. Planned concurrent surgical procedure with the exception of salpingo-oophorectomy or tubal ligation.
4. Use of any of the following medications within the times specified before surgery: long-acting opioid medication, non-steroidal anti-inflammatory drugs (NSAIDs), or aspirin (except for low-dose aspirin used for cardioprotection) within 3 days, or any opioid medication or acetaminophen within 24 hours.
5. Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®). If a subject is taking one of these medications for a reason other than pain control, she must be on a stable dose for at least 1 month prior to study drug administration.
6. Clinically significant medical or psychiatric disease that, in the opinion of the Investigator, would constitute a contraindication to participation in the study or cause inability to comply with the study requirements.
7. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medication(s), or alcohol within the past 2 years.
8. Received an investigational drug within 30 days prior to study drug administration, and/or has planned administration of another investigational product or procedure while participating in this study.
9. Previous participating in an EXPAREL study.

   The subject will be withdrawn from the study if she meets the following criteria:
10. Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postsurgical course.
11. Her baby's 5-minute Apgar score is ≤7.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erol Onel, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (5):
- United States (5):
  - Tradition Medical Center, Port Saint Lucie, Florida
  - University Of Minnesota, Minneapolis, Minnesota
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Montefiore, The Bronx, New York
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | EXPAREL/TAP
Started | 12 | 0
Completed | 10 | 0
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated due to slow enrollment after 12 subjects were assigned to Group 1 (Standard of Care/Duramorph). As no subjects were enrolled into Group 2 (EXPAREL/TAP), no conclusions can be drawn regarding the study endpoints.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | EXPAREL/TAP | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 12 |  | 12
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (4.71) |  | 32.2 (4.71)
Sex/Gender, Customized [Number; unit: participants]
  Female | 12 |  | 12
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Total Postsurgical Narcotic Consumption in Morphine Equivalents
Description: Outcome measure data refer to 7 participants who received rescue medication
Time Frame: Through 72 hours postdose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: MUEs
Arm/Group | Standard of Care | EXPAREL/TAP
Number analyzed (Participants) | 12 | 0
MUEs | 6.1 (3.67) |

2. Secondary Outcome: Total Postsurgical Narcotic Consumption in Morphine Equivalents
Description: Outcome measure data refer to 6 participants who received rescue medication
Time Frame: Through 24 hours
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: MUEs
Arm/Group | Standard of Care | EXPAREL/TAP
Number analyzed (Participants) | 12 | 0
MUEs | 4.9 (2.01) |

3. Secondary Outcome: Total Postsurgical Narcotic Consumption in Morphine Equivalents
Description: Outcome measure data refer to 7 participants who received rescue medication
Time Frame: Through 48 hours
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: MUEs
Arm/Group | Standard of Care | EXPAREL/TAP
Number analyzed (Participants) | 12 | 0
MUEs | 6.1 (3.67) |

ADVERSE EVENTS:
Arm/Group | Standard of Care | EXPAREL/TAP
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/0
Other Adverse Events (participants affected / at risk) | 2/12 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=12) | EXPAREL/TAP (N=0)
oral herpes (Infections and infestations) | 1 (1) | 0 (0)
bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No